CLINICAL TRIAL: NCT03888300
Title: VLM-2: Measurement of Viscoelastic Properties of Bronchopulmonary Secretions.
Brief Title: Measurement of Viscoelastic Properties of Bronchopulmonary Secretions.
Acronym: VLM-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/17OCT/391
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: All patients will receive standard physiotherapy as prescribed by the physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Group (Experimental): Patients with obstructive pulmonary diseases receiving standard physiotherapy treatment
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Chest Physiotherapy, physical exercises

SUMMARY:
The study is experimental and aims to (a) compare the viscoelastic properties of bronchial secretions obtained in patients suffering from obstructive respiratory disease, and (b) to compare the viscoelastic properties of bronchial secretions obtained in patients before and after application of a respiratory physiotherapy or exercise as usually prescribed.

After agreement, the sputum of the participants will be collected according to the method used in clinical routine.Experiments (collection and analysis of sputum) will be conducted at the Saint-Luc University Clinic.

ELIGIBILITY:
Inclusion Criteria:

* obstructive pulmonary disease

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Viscoelasticity | 30 minutes
  Evolution of elastic modulus, viscous modulus, phase angle and non-linear characteristics of lung secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reychler, PT, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No